CLINICAL TRIAL: NCT07363564
Title: The Prevalence of Hand Joint Hypermobility and Its Relationship With Grip Strength Among University Students
Status: Not yet recruiting | Type: Observational
Sponsor: Ehab A. Abdallah (Other)
Collaborators: Horus University (Other)
Responsible Party: Sponsor-Investigator, Ehab A. Abdallah, ASSOCIATE PROFESSOR, Horus University
Organization: Horus University (Other)
Other Study IDs: (Approval No: P.T.REC/012/0047
Record Dates: First submitted 2026-01-05; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hand Joint Hypermobility; Grip Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Interventions — NO INTERVENTION

SUMMARY:
This cross-sectional study investigated the prevalence of hand joint hypermobility among 400 university students and its relationship with hand grip strength. MCP joint mobility was assessed using a universal goniometer, and grip strength was measured with a hand dynamometer. Participants were categorized into mild, moderate, and severe hypermobility groups.

DETAILED DESCRIPTION:
Objective: This study aims to determine the prevalence of hand joint hypermobility among university students and examine its association with hand grip strength. Specifically, it seeks to compare grip strength between students with and without hypermobility and explore potential implications for educational activities such as writing and studying.

Design: A descriptive cross-sectional study was conducted among 400 students. Settings: 400 students recruited from both public and private universities. Participants: Students were assessed at the metacarpophalangeal (MCP) joints using a universal goniometer, while hand grip strength was measured with an adjustable hand dynamometer. Based on MCP range of motion, participants were categorized into three groups: mild, moderate, and severe hypermobility.

Intervention: Not Applicable. Main outcome measures: Metacarpophalangeal (MCP) joint hypermobility was measured using a universal goniometer, and grip strength was assessed using a hand dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible if they were undergraduate university students enrolled in the 2023/2024 academic year, male or female, aged between 18 and 22 years, and had no previously diagnosed systemic conditions associated with hypermobility (e.g., Ehlers-Danlos syndrome or generalized hypermobility syndrome).

Exclusion Criteria:

* Participants were excluded if they had a previously diagnosed systemic condition associated with hypermobility, reported musculoskeletal injuries or conditions affecting joint mobility or grip strength at the time of assessment, were unable or unwilling to provide informed consent, had any neurological or chronic disorders that could influence muscle strength or joint range of motion or were outside the specified age range (18-22 years).

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 400 male and female students aged 18-22 years were recruited from multiple universities to ensure diversity and representativeness. The sample included students from public institutions and a private institution. This multi-center approach was designed to capture variability in demographics and educational environments
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Metacarpophalangeal (MCP) joint hypermobility was measured using a universal goniometer, | 1 JAN 2026 TO 30 JAN 2026
grip strength was assessed using a hand dynamometer | once
  and grip strength was assessed using a hand dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Horus University, Damietta, Da, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Remvig L, Jensen DV, Ward RC. Epidemiology of general joint hypermobility and basis for the proposed criteria for benign joint hypermobility syndrome: review of the literature. J Rheumatol. 2007 Apr;34(4):804-9. Epub 2007 Jan 15. PMID 17407233

DOCUMENTS (1):
  • Study Protocol (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT07363564/Prot_000.pdf